CLINICAL TRIAL: NCT06817863
Title: A Self-Guided Mobile Intervention for Adults With Binge Eating and Obesity
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Oui Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2408010718; R41MH134704 (NIH)
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Binge Eating Disorder Associated With Obesity; Binge Eating Disorder
Keywords: digital treatment; self-help intervention; binge eating
MeSH Terms: conditions — Binge-Eating Disorder; Bulimia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-Help Digital Intervention (Experimental): All study participants will receive the digital intervention (ChangeBite). Therefore, this study has 1 arm.
  Interventions: Other: Digital

INTERVENTIONS:
Other: Digital — This intervention is a self-help digital treatment, delivered via a smartphone application, for adults with co-morbid binge eating and obesity. The app ChangeBite will integrate principles of evidence based treatments for obesity (behavioral weight loss treatment) and binge eating (cognitive behavioral therapy, acceptance and commitment therapy) into a highly personalized, self-guided, program that leverages an artificial conversational agent and Just-In-Time-Adaptive-Interventions (JITAIs).

SUMMARY:
The proposed study is an open label, non randomized, waitlist controlled single group feasibility study of the feasibility and usability of a digital intervention (called ChangeBite) to be used by individuals with obesity and comorbid binge eating behavior. The proposed research will include approximately 30 participants. Participants will be recruited for this single group pilot trial using online advertising to attend a virtual screening session. Screened participants willing and eligible to participate, will receive informed consent and formally start ChangeBite. Participants will be instructed to engage with ChangeBite and attend follow up assessments on scheduled video calls. Feasibility and acceptability of implementation will be assessed by collecting data on recruitment, retention, usability and satisfaction. The research team will also collect assessment data from participants on feasibility, and usability. In addition to self report scales, semi-structured interviews will be completed with a trained research team member via video call and will be partially recorded. Assessments will be done at baseline, 12 weeks, and 24 weeks. Participants' app use frequency and duration will be tracked using software analytics. Participants' body weight will be captured weekly using a timestamped picture of their weight as it appears on their scale and Body Mass Index will be calculated with these data points.

ELIGIBILITY:
Inclusion Criteria:

1. Are English speaking male or female
2. Are aged 18-70 years
3. Have recurrent objective or subjective binge eating episodes (≥12 episodes in 3 months)
4. Have BMI ≥30
5. Own an iPhone with iOS 11 or higher, or Android with OS 8.1 or higher
6. Are willing and able to complete enrollment procedures
7. Are able to understand the nature of the study and provide written informed consent

Exclusion Criteria:

1. Are unable to fluently speak, write and read English.
2. Are already receiving treatment for an eating disorder (e.g., research participants cannot be receiving concurrent eating disorder treatment from another provider)
3. Are receiving weight loss treatment (behavioral or pharmacological)
4. Have a mental handicap or are currently experiencing severe psychopathology that would limit their ability to engage in study (e.g., imminent or high risk for suicide, substance use disorder, active psychotic disorder,)
5. Are purging and/or using laxatives 3 or more times per week and are not deemed safe for remote treatment by a primary care provider.
6. Are exercising 2 or more hours a day on average, or engaging in significantly harmful compensatory behaviors (i.e., > 3x/week of self-induced vomiting or laxative use), and are not deemed safe for remote treatment by a primary care provider.
7. Are fasting for 24 hours or more, > 3x times a week, and are not deemed safe for remote treatment by a primary care provider.
8. Are unwilling to receive medical clearance and/or medical monitoring as requested by the study to ensure they are medically safe to participate.
9. Are pregnant or planning to become pregnant within the next year.
10. Are individuals who are not yet adults (infants, children, teenagers) Are currently taking any of these medications: Haldol, Loxitane, Mellaril, Moban, Navane, Prolixin, Serentil, Stelaxine, Trilafon, Thoraxine, Abilify, Clozaril, Geodon, Risperdal, Seroquel, Zyprexa
11. Are adults unable to consent
12. Are prisoners

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Binge eating episodes | 3 months
  The frequency of binge eating episodes.
Weight | 3 months
  Weight loss during the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes